CLINICAL TRIAL: NCT03078335
Title: Non-Sterile Glove Based Care to Prevent Late Onset Sepsis in The NICU - Cluster Crossover Randomized Controlled Pilot Study
Brief Title: Glove-based Care in the NICU to Prevent Late Onset Sepsis
Acronym: GloveCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GloveCare
Record Dates: First submitted 2017-02-01; First posted 2017-03-13 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Sepsis Newborn; Infection
Keywords: Late onset sepsis; glove based care; NICU; Non sterile gloves; infection control
MeSH Terms: conditions — Neonatal Sepsis; Infections

STUDY DESIGN:
Intervention Model Description: This pilot study is a single centre NICU based cluster-randomized crossover trial, with 2 crossover periods each lasting 6 months, and a 2-week washout period in between.
Who Masked: Outcomes Assessor
Masking Description: The final adjudication of events will be completed by two of the investigators blinded to study arm, based on a summary report of each event after completion of the pilot.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glove based care (Experimental): The intervention is the use of non-sterile gloves, after standard hand hygiene for all routine patient care needs.
  Interventions: Other: Glove based care
- Standard care (Active Comparator): The control group will provide standard care, that is, hand hygiene before all patient, bed, and intravenous catheter contact.
  Interventions: Other: Standard of Care - Hand Hygiene

INTERVENTIONS:
Other: Glove based care — Described in Experimental Arm: Glove based care
  Arms: Glove based care
Other: Standard of Care - Hand Hygiene — Hand Hygiene - hand washing with soap and water, or alcohol based hand rub
  Arms: Standard care

SUMMARY:
Babies that get an infection after 3 days of age while in the Neonatal Intensive Care Unit is not related to their delivery but to the hospital environment. Preventing these infections results in shorter hospital stays for babies, less risk of long term health problems and less health care resources required to care for them. Hand washing alone doesn't remove all bacteria from the hands of healthcare workers, and studies have shown that infections in adults and children admitted to hospital decrease if health care providers use clean, non- sterile gloves when treating patients. The main focus of this study will be to find out if using gloves when caring for newborns in the NICU is better than washing hands alone. McMaster Children's Hospital and The Hospital for Sick Children will be the pilot sites to participate in a future larger study where some infants will be cared for using non-sterile gloves, and others will be cared for using the standard hand washing method.

DETAILED DESCRIPTION:
Late onset sepsis (LOS) is defined as infection occurring after 72 hours of life in neonates admitted to the Neonatal Intensive Care Unit (NICU). LOS can lead to severe complications including death, major neurologic sequelae, and contribute to increased length of stay and costs of care. These hospital acquired infections are largely preventable. Hand washing prior to any patient care is considered the cornerstone of prevention and is the standard of care in the NICU. Adherence to hand washing however is difficult to achieve, with estimates of compliance among health care workers ranging from 30% to 60%. Observational studies in at-risk critically ill children suggest a reduction in hospital acquired infections and central line associated bloodstream infections with glove based care in addition to hand hygiene. One small single-centre randomized trial of glove based care versus hand hygiene alone to assess LOS rates in extremely premature infants in the NICU showed a reduction in gram positive infections and central line infections with glove-based care. We propose to test the effect of glove based care in an adequately powered, rigorously designed and conducted, cluster randomized controlled trial (RCT) after completing a feasibility pilot study.

This pilot study will include all babies in the NICU being randomized to 6 months of glove based care or standard of care, and then the following 6 months will be the opposite arm. All health care provider contact with the infant will require gloves in the intervention arm, but families of infants admitted to the NICU will not be required to wear gloves. The main outcome measured will be the number of episodes of infections in the blood, urinary tract, and cerebrospinal fluid comparing the glove intervention arm against the control arm. Invasive infections are an important challenge for infants admitted to the NICU and reducing this risk can improve the quality and quantity of neonatal survivors from the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the NICU at participating sites for > 2 days until discharge

Exclusion Criteria:

* Babies requiring contact precautions due to other reasons (as glove based care would be occurring)

Min Age: 1 Minute | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 786 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Late onset sepsis events | Weeks of admission to the NICU. Infection must occur at >72 hours of age, throughout neonatal admissions for the 6 month duration of each study arm
  The anticipated incidence of LOS is 10% of patients based on Canadian Neonatal Network retrospective data. Infection is defined as blood stream, urinary tract, or cerebrospinal fluid infection based on 1 or more positive cultures with a bacterial or fungal pathogen (2 cultures required for Coagulase negative staphylococcus), at least 2 compatible signs and symptoms (including temperature instability, hemodynamic changes, respiratory distress and increased inflammatory markers), and the need for antimicrobial treatment.

SECONDARY OUTCOMES:
Time to first infection | Time from admission to NICU to discharge (days to months) throughout neonatal admissions for the 6 month duration of each study arm]
  Time from admission to NICU to first infection in days
Length of stay | Time from admission to discharge (days to months) throughout neonatal admissions for the 6 month duration of each study arm]
  Time from admission to discharge (days)
All-cause mortality | Duration of study (1 year)
  Number of deaths (number of patients who die during study)
Proportion colonized by antibiotic resistant organisms at any point during their NICU stay | Weeks of admission to NICU, for the duration of study (1 year)
  Proportion of infants who become colonized with antibiotic resistant organisms during surveillance screening as part of routine care (number of patients)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Khan, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoll BJ, Hansen NI, Bell EF, Walsh MC, Carlo WA, Shankaran S, Laptook AR, Sanchez PJ, Van Meurs KP, Wyckoff M, Das A, Hale EC, Ball MB, Newman NS, Schibler K, Poindexter BB, Kennedy KA, Cotten CM, Watterberg KL, D'Angio CT, DeMauro SB, Truog WE, Devaskar U, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Trends in Care Practices, Morbidity, and Mortality of Extremely Preterm Neonates, 1993-2012. JAMA. 2015 Sep 8;314(10):1039-51. doi: 10.1001/jama.2015.10244. PMID 26348753
- [Background] Orcesi S, Olivieri I, Longo S, Perotti G, La Piana R, Tinelli C, Spinillo A, Balottin U, Stronati M. Neurodevelopmental outcome of preterm very low birth weight infants born from 2005 to 2007. Eur J Paediatr Neurol. 2012 Nov;16(6):716-23. doi: 10.1016/j.ejpn.2012.05.006. Epub 2012 Jun 17. PMID 22709626
- [Background] Alemagno SA, Guten SM, Warthman S, Young E, Mackay DS. Online learning to improve hand hygiene knowledge and compliance among health care workers. J Contin Educ Nurs. 2010 Oct;41(10):463-71. doi: 10.3928/00220124-20100610-06. Epub 2010 Jun 8. PMID 20540459
- [Background] Yin J, Schweizer ML, Herwaldt LA, Pottinger JM, Perencevich EN. Benefits of universal gloving on hospital-acquired infections in acute care pediatric units. Pediatrics. 2013 May;131(5):e1515-20. doi: 10.1542/peds.2012-3389. Epub 2013 Apr 22. PMID 23610206
- [Background] Johnson S, Gerding DN, Olson MM, Weiler MD, Hughes RA, Clabots CR, Peterson LR. Prospective, controlled study of vinyl glove use to interrupt Clostridium difficile nosocomial transmission. Am J Med. 1990 Feb;88(2):137-40. doi: 10.1016/0002-9343(90)90462-m. PMID 2301439
- [Background] Kaufman DA, Blackman A, Conaway MR, Sinkin RA. Nonsterile glove use in addition to hand hygiene to prevent late-onset infection in preterm infants: randomized clinical trial. JAMA Pediatr. 2014 Oct;168(10):909-16. doi: 10.1001/jamapediatrics.2014.953. PMID 25111196
- [Background] Edwards WH, Conner JM, Soll RF; Vermont Oxford Network Neonatal Skin Care Study Group. The effect of prophylactic ointment therapy on nosocomial sepsis rates and skin integrity in infants with birth weights of 501 to 1000 g. Pediatrics. 2004 May;113(5):1195-203. doi: 10.1542/peds.113.5.1195. PMID 15121929
- [Background] Shah J, Jefferies AL, Yoon EW, Lee SK, Shah PS; Canadian Neonatal Network. Risk Factors and Outcomes of Late-Onset Bacterial Sepsis in Preterm Neonates Born at < 32 Weeks' Gestation. Am J Perinatol. 2015 Jun;32(7):675-82. doi: 10.1055/s-0034-1393936. Epub 2014 Dec 8. PMID 25486288
- [Background] Tsai MH, Hsu JF, Chu SM, Lien R, Huang HR, Chiang MC, Fu RH, Lee CW, Huang YC. Incidence, clinical characteristics and risk factors for adverse outcome in neonates with late-onset sepsis. Pediatr Infect Dis J. 2014 Jan;33(1):e7-e13. doi: 10.1097/INF.0b013e3182a72ee0. PMID 23899966
- [Background] Samuelsson A, Isaksson B, Hanberger H, Olhager E. Late-onset neonatal sepsis, risk factors and interventions: an analysis of recurrent outbreaks of Serratia marcescens, 2006-2011. J Hosp Infect. 2014 Jan;86(1):57-63. doi: 10.1016/j.jhin.2013.09.017. Epub 2013 Oct 23. PMID 24332914
- [Background] Dong Y, Speer CP. Late-onset neonatal sepsis: recent developments. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F257-63. doi: 10.1136/archdischild-2014-306213. Epub 2014 Nov 25. PMID 25425653
- [Background] Wong JL, Siti Azrin AH, Narizan MI, Norliah Y, Noraida M, Amanina A, Nabilah I, Habsah H, Siti Asma H. Back to basic: bio-burden on hands of health care personnel in tertiary teaching hospital in Malaysia. Trop Biomed. 2014 Sep;31(3):534-9. PMID 25382481
- [Background] Sharma VS, Dutta S, Taneja N, Narang A. Comparing hand hygiene measures in a neonatal ICU: a randomized crossover trial. Indian Pediatr. 2013 Oct;50(10):917-21. doi: 10.1007/s13312-013-0261-3. Epub 2013 Mar 5. PMID 23585422
- [Background] Monistrol O, Lopez ML, Riera M, Font R, Nicolas C, Escobar MA, Freixas N, Garau J, Calbo E. Hand contamination during routine care in medical wards: the role of hand hygiene compliance. J Med Microbiol. 2013 Apr;62(Pt 4):623-629. doi: 10.1099/jmm.0.050328-0. Epub 2013 Jan 17. PMID 23329322
- [Background] Moolenaar RL, Crutcher JM, San Joaquin VH, Sewell LV, Hutwagner LC, Carson LA, Robison DA, Smithee LM, Jarvis WR. A prolonged outbreak of Pseudomonas aeruginosa in a neonatal intensive care unit: did staff fingernails play a role in disease transmission? Infect Control Hosp Epidemiol. 2000 Feb;21(2):80-5. doi: 10.1086/501739. PMID 10697282
- [Background] Jefferies JMC, Cooper T, Yam T, Clarke SC. Pseudomonas aeruginosa outbreaks in the neonatal intensive care unit--a systematic review of risk factors and environmental sources. J Med Microbiol. 2012 Aug;61(Pt 8):1052-1061. doi: 10.1099/jmm.0.044818-0. Epub 2012 Jun 8. PMID 22683659
- [Background] Coffin SE. Fighting infections in the neonatal intensive care unit: gloves on or off? JAMA Pediatr. 2014 Oct;168(10):885-7. doi: 10.1001/jamapediatrics.2014.1269. No abstract available. PMID 25111036
- [Background] Harris AD, Pineles L, Belton B, Johnson JK, Shardell M, Loeb M, Newhouse R, Dembry L, Braun B, Perencevich EN, Hall KK, Morgan DJ; Benefits of Universal Glove and Gown (BUGG) Investigators; Shahryar SK, Price CS, Gadbaw JJ, Drees M, Kett DH, Munoz-Price LS, Jacob JT, Herwaldt LA, Sulis CA, Yokoe DS, Maragakis L, Lissauer ME, Zervos MJ, Warren DK, Carver RL, Anderson DJ, Calfee DP, Bowling JE, Safdar N. Universal glove and gown use and acquisition of antibiotic-resistant bacteria in the ICU: a randomized trial. JAMA. 2013 Oct 16;310(15):1571-80. doi: 10.1001/jama.2013.277815. PMID 24097234
- [Background] Klein BS, Perloff WH, Maki DG. Reduction of nosocomial infection during pediatric intensive care by protective isolation. N Engl J Med. 1989 Jun 29;320(26):1714-21. doi: 10.1056/NEJM198906293202603. PMID 2733733
- [Background] Tan SG, Lim SH, Malathi I. Does routine gowning reduce nosocomial infection and mortality rates in a neonatal nursery? A Singapore experience. Int J Nurs Pract. 1995 Nov;1(1):52-8. doi: 10.1111/j.1440-172x.1995.tb00009.x. PMID 9264888
- [Derived] Khan S, Tsang KK, Hu ZJ, Mostowiak B, El Helou S, Science M, Kaufman D, Pernica J, Thabane L, Mertz D, Loeb M. GloveCare: a pilot study in preparation for a cluster crossover randomized controlled trial of non-sterile glove-based care in preventing late-onset infection in the NICU. Pilot Feasibility Stud. 2023 Mar 23;9(1):50. doi: 10.1186/s40814-023-01271-9. PMID 36959636